CLINICAL TRIAL: NCT03678389
Title: Feasibility of Endosphenoidal Coil Placement for Imaging of the Sella During Transsphenoidal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 180133; 18-N-0133
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-06-17

CONDITIONS: Pituitary Neoplasm
Keywords: Pituitary Adenoma; pituitary surgery; Transsphenoidal Surgery; Pituitary Tumors
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): ENDOSPHENOIDAL COIL
  Interventions: Other: ESC

INTERVENTIONS:
Other: ESC — USE OF ENDOSPHENOIDAL COIL (ESC) TO OBTAIN MRI IMAGING OF THE PITUITARY GLAND

SUMMARY:
Background:

Pituitary tumors can cause problems by secreting hormones in the body. They can also problems by growing large and pushing on organs near the pituitary gland. The best treatment for such tumors is to remove them by surgery. But that may be sometimes difficult. Some tumors maybe too small to see. Some other tumors maybe so large that portions maybe left behind during surgery. The endosphenoidal coil (ESC) is a new magnetic resonance imaging (MRI) device. It fits in a small space made during surgery near the pituitary. Researchers want to see if it helps transmit MRI signals during surgery to make better images of the pituitary gland and tumors.

Objective:

To test the safety of using a new coil device to improve MRI imaging of pituitary tumors during surgery.

Eligibility:

Adults 18-85 years old who are having pituitary tumor surgery at NIH

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Review of prior brain scans
* Blood and pregnancy tests

All participants will have MRI of pituitary gland. They will lie on a table that slides into a metal cylinder in a strong magnetic field. They will lie still and get earplugs for loud sounds. A dye will be inserted into an arm vein by needle.

Participants will stay in the hospital for about 1 week. They will repeat screening tests.

Participants will have standard pituitary surgery. They will get medicine to go to sleep. The surgeon will create a path to the pituitary gland from under the lip.

During surgery, the ESC will be placed through the path to near the pituitary. Then an MRI will be done during surgery.

Then the ESC will be removed and standard surgery will continue.

Participants will get standard post-operative care under another protocol....

DETAILED DESCRIPTION:
Tumors of the pituitary gland comprise up to 20% of all brain tumors. The central location and the small size of the pituitary gland make the management of tumors particularly challenging. Transsphenoidal surgery (TSS) to resect pituitary tumors is highly successful at achieving a complete cure for functional pituitary adenomas. It is most successful when such adenomas can be localized by preoperative MRI of the pituitary. However, in some instances, small functional tumors cannot be visualized. In the case of Cushing s disease (CD), such non-visualization may be as high as 50%. The success of transsphenoidal surgery is substantially reduced in patients with negative MRI, as some of the adenomas that cause CD are so small that they are difficult to find during surgical exploration of the pituitary. Surgical success is also diminished when tumors invade the walls of the cavernous sinus. MRI of the pituitary lacks imaging resolution to detect such invasion, so the surgeon cannot perform a complete resection with surgery based on the preoperative MRI.

Signal-to-noise ratio (SNR) is the primary constraint on achieving high-quality high-resolution MRI images. SNR can be improved by longer scan times or by increasing the field strength of the MRI magnet. SNR is proportional to the square of imaging time. However, long imaging times are not clinically feasible. SNR is linearly proportional to field strength. However, replacing MRI magnets is cost- prohibitive.

Another strong determinant of SNR is the proximity of the MRI receiver coil to the tissue being imaged. Placement of a coil in close proximity to the structure of interest dramatically increases SNR, often as much as 10-fold. Clinically this is routinely put into practice for superficial body parts, such as the temporomandibular joints, in which small coils are placed directly over the joints to achieve rapid high-resolution imaging. For deep structures, the use of superficial coils is of no benefit. This has led to the development of endocavitary coils, such as the endorectal coil used to image the prostate gland. Such coils are now in routine clinical use here at the NIH and elsewhere.

During routine TSS, the surgical approach to the pituitary gland provides a route for the placement of imaging tools, such as handheld ultrasound and Doppler probes in close proximity to the gland. Extending this model to MRI imaging, we realized that an endocavitary surface coil within the sphenoid sinus would allow for a marked improvement in SNR for imaging the sella. To this end, we have developed an endosphenoidal coil (ESC), demonstrated its MRI safety, and performed preliminary studies in cadaver heads to determine that the ESC can be placed through the transsphenoidal approach. The placement of ESC needs no modification in the surgical TSS approach to the pituitary gland. The goal of this protocol is to examine the safety and feasibility of ESC placement and imaging during TSS.

Objective

To evaluate the feasibility and safety of using ESC during TSS.

Study Population

The study population will be up to 70 adult subjects with pituitary tumors that require TSS. Enrollment will be completed once 50 subjects have received the study procedure. The requested accrual ceiling of 70 subjects accounts for screening failures and drop-outs who do not receive the study procedure.

Design

This is a pilot study of 50 subjects requiring TSS for pituitary lesions. The subjects will undergo standard TSS resection of a pituitary adenoma in the intra-operative MR suite. Following the standard surgical approach, the ESC will be placed into the sphenoid sinus while the bone of the sellar floor is still intact. Routine clinical pituitary imaging with and without intravenous contrast will be performed for comparison with standard pituitary imaging. Additional higher-resolution sequences will be performed as time allows. Following imaging, standard surgical resection will be performed. The surgeon will not view scans arising from the research procedure, and therefore intraoperative clinical decision-making will not be influenced by the results of the research imaging.

Outcome Measures:

Primary Outcome Measure

Preliminary analysis of the data generated so far revealed that the ESC is well-designed to fit within the surgical workflow. However, the utility of ESC imaging was limited within the parameters of the standard sequences. Depending on the specific clinical indication for TSS, we found that the ESC could have differing roles as a surgical adjunct. For the current amended trial, the feasibility of ESC will be evaluated as follows:

1. For microadenomas (pituitary adenomas smaller than 10 mm in diameter), the ability of ESC to confirm the location and size of adenomas.
2. For macroadenomas (pituitary adenomas larger than 10 mm in diameter), the ability of ESC to detect invasion of the cavernous sinus and/or parasellar structures (structures surrounding the pituitary gland).
3. For MRI-negative cases, the ability to detect adenomas.

Safety Outcome Measure

We will evaluate the safety of the ESC as a surgical adjunct tool. We will evaluate whether the use of ESC causes local trauma, bleeding, burns or other unanticipated safety issues during TSS.

Exploratory Outcome Measures

Clinical utility of these images will be evaluated by comparing SNR and contrast to noise ratio (CNR) measurements obtained with the ESC to preoperative standard of care images.

1. Pituitary SNR with ESC MRI versus pre-operative standard of care images.
2. Pituitary to tumor Contrast to Noise Ratio (CNR) with ESC MRI versus pre-operative standard of care images.

ELIGIBILITY:
* INCLUSION CRITIERIA:

Adult subjects (more than 18 years of age) will be included in this study if they:

1. Have a known or suspected tumor of the pituitary gland that requires surgical resection through a transsphenoidal approach. There is no size restriction. Invasion of surrounding anatomical structures by the pituitary tumor will not be ground for screen failure/withdrawal from study.
2. Are enrolled in 03-N-0164, Evaluation and Treatment of Neurosurgical Disorders. If not enrolled, subjects will not be able to be included in the study as clinical and research procedures are done under the 03-N-0164 protocol.
3. Are able to provide written consent.
4. NIH employees are included in the study.

EXCLUSION CRITIERIA:

Subjects will be excluded from this study if they:

1. Are unable to fit the intra-operative MRI table due to size or weight restrictions i.e morbid obesity. Patients will be anaesthetized and therefore claustrophobia will not be ground for screen failure/withdrawal from study.
2. Have an absolute contraindication to MRI imaging or MRI contrast agent according to Rad&IS screening including devices or conditions.
3. Have a variant anatomy which may, in the judgment of the operating neurosurgeon, add unacceptable risk to the placement of the endosphenoidal coil (e.g. small size of facial bones and nasal passages, unaerated sphenoid sinus etc.).
4. Are pregnant or nursing.
5. Patients older than 85 years of age. Cushing disease is rare in the older population.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using ESC as a clinical tool during transsphenoidal surgery. Feasibility will be assessed by the time added to a standard TSS procedure. | 2 hours
  The primary outcome of this study is the feasibility of using ESC as a clinical tool during transsphenoidal surgery. Feasibility will be assessed by the time added to a standard TSS procedure (measured from the time the TSS exposure is completed to the time to return to the operating position for completion of surgery).

SECONDARY OUTCOMES:
Evaluate whether the use of ESC causes local trauma, bleeding, burns or other unanticipated safety issues during TSS. | Study Completion

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Chittiboina, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do plan to share IPD. We will share all IPD that results in a publication on a public repository, as required by most journals. The data will be de-identified and anonymized.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-N-0133.html